CLINICAL TRIAL: NCT07003698
Title: Postoperative Analgesic Efficacy of Rectointercostal Nerve Block in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Postoperative Analgesic Efficacy of Recto Intercostal Nerve Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Muruvvet Taskir Turan, Principal investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-009
Record Dates: First submitted 2025-04-10; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Laparoskopic Cholecystectomy; Recto Intercostal Nerve Block
Keywords: Remifantanile conception; Acute pain; Postoperatif pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group without rectointercostal nerve block (Active Comparator): Patients in this group will be administered dexketoprofen 50 mg and tramadol 100 mg intravenously in the intraoperative period. These patients will not receive the rectointercostal nerve block.
  Interventions: Procedure: The group without the rectointercostal nerve block
- Postoperative analgesic efficacy of rectointercostal nerve block (Active Comparator): The patient lies in the supine position. The skin is disinfected. A high-frequency linear probe (6-13 MHz) is placed lateral to the xiphoid to visualize the rectus abdominis muscle at the level of the 7th rib. Using an in-plane technique, a 22G, 80 mm block needle is inserted in a cranial direction into the interfascial plane immediately inferolateral to the xiphoid, between the rectus abdominis muscle and the 6th-7th costal cartilages. A total of 20 ml of local anesthetic solution is injected bilaterally (40 ml of 0.25% bupivacaine (marcaine)). The spread of the local anesthetic is confirmed by ultrasound guidance.
  Additionally, patients in this group will be administered dexketoprofen 50 mg and tramadol 100 mg intravenously in the intraoperative period.
  Interventions: Procedure: The rectointercostal plane block

INTERVENTIONS:
Procedure: The group without the rectointercostal nerve block — Patients in this group will be administered dexketoprofen 50 mg and tramadol 100 mg intravenously in the intraoperative period. These patients will not receive the rectointercostal nerve block.
  Arms: The group without rectointercostal nerve block
Procedure: The rectointercostal plane block — The rectointercostal plane block is performed under ultrasound guidance before the surgical procedure and anesthesia induction, with the patient in the supine position. Additionally, patients in this group will be administered dexketoprofen 50 mg and tramadol 100 mg intravenously in the intraoperative period.
  Arms: Postoperative analgesic efficacy of rectointercostal nerve block

SUMMARY:
Laparoscopic cholecystectomy is a frequently performed surgery and the gold standard for the treatment of symptomatic gallstone disease. Although laparoscopic cholecystectomy is considered minimally invasive, it can cause moderate to severe pain in the postoperative period. Poorly controlled early postoperative pain impairs recovery quality and increases the risk of postoperative pulmonary complications, serving as a risk factor for chronic pain development.

Multimodal analgesia, including opioids, is used to manage pain following laparoscopic cholecystectomy. However, opioid treatment may lead to side effects such as postoperative nausea and vomiting (PONV), respiratory depression, and constipation.

The primary aim of this study is to evaluate the effect of recto-intercostal nerve block as part of multimodal analgesia on intraoperative opioid consumption and postoperative pain scores in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* Elective laparoscopic cholecystectomy surgery

Exclusion Criteria:

* Under 18 and over 65 years old
* ASA score IV and above
* Advanced co-morbidity
* History of bleeding diathesis
* Patient refusing the procedure
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Block injection site infection
* Known allergy to local anesthetics
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-22 (Estimated); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption | During the intraoperative period
  The amount of remifentanil that patients need to maintain anesthesia during the intraoperative period will be recorded

SECONDARY OUTCOMES:
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while movement using the from 0 (no pain) to 10 (worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)